CLINICAL TRIAL: NCT01581216
Title: The Use of Physical Activity to Control Fatigue and Improve the Quality of Life in Patients With Advanced Cancer Stage
Brief Title: Fatigue Before and After Exercise in Patients With Advanced Cancer Stage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Barretos Cancer Hospital (Other)
Responsible Party: Principal Investigator, Adriana Silva Martins Ferreira, Principal Investigator, Barretos Cancer Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: fatigue-hcb-01
Record Dates: First submitted 2012-02-01; First posted 2012-04-20 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-08

CONDITIONS: Fatigue
Keywords: Fatigue; Palliative Care; Exercise
MeSH Terms: conditions — Fatigue; Motor Activity | interventions — Walking; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 10 minute walk (Experimental): 10-minute walk and exercises for the upper limbs with 1 lb-dumbbells
  Interventions: Other: 10 minute walk
- 20 minute walk (Experimental): 20-minute walk and exercises for the upper limbs with 1 lb-dumbbells
  Interventions: Other: 20 minute walk
- 30 minute walk (Experimental): 30-minute walk and exercises for the upper limbs with 1 lb-dumbbells
  Interventions: Other: 30 minute walk

INTERVENTIONS:
Other: 10 minute walk — Patients who walk a distance ≤ 300 meters in the 6-minute walk test will make a 10 minute walk once a day for 5 days for 4 weeks in a 90-feet long corridor located at the palliative care unit.
  Other Names: 10 minute walk and exercises
  Arms: 10 minute walk
Other: 20 minute walk — Patients who walk 300-450 meters in the 6-minute walk test will make a 20 minute walk once a day for 5 days for 4 weeks in a 90-feet long corridor located at the palliative care unit.
  Other Names: 20 minute walk and exercises
  Arms: 20 minute walk
Other: 30 minute walk — Patients who walk a distance less than 450 meters in the 6-minute walk test will make a 30 minute walk once a day for 5 days for 4 weeks in a 90-feet long corridor located at the palliative care unit.
  Other Names: 30 minute walk and exercises
  Arms: 30 minute walk

SUMMARY:
Fatigue related to cancer is the most common reported symptom and it prevents 91% of patients of having an active life, and in several cases, the fatigue persists for several months or even years after treatment. Fatigue does cause an impact in all dimensions of patients' quality of life and it is the main cause of reduction in patients' daily life activities.

Fatigue is reported by cancer patients in all phases of the illness as one of the most frequent symptoms, especially in cases presenting metastases.

In order to monitor fatigue, pharmacological and non-pharmacological techniques may be employed, such as physical activity. Physical exercise has shown positive results in mitigating fatigue improving cardiopulmonary functioning, physical capacity and patients' quality of life.

This study will assess the efficiency of physical activity upon controlling the fatigue and quality of life in patients with advanced stage of the disease at the end of 7 days using FACT-F subscale.

DETAILED DESCRIPTION:
Six minute walking test: a) Patients who walk a distance ≤ 300 meters in the 6-minute walk test will make a 10 minute walk once a day for 5 days for 4 weeks in a 30-feet long corridor located at the palliative care unit; b) Patients who walk 300-450 meters in the 6-minute walk test will make a 20 minute walk once a day for 5 days for 4 weeks in a 30-feet long corridor located at the palliative care unit; c) Patients who walk a distance less than 450 meters in the 6-minute walk test will make a 30 minute walk once a day for 5 days for 4 weeks in a 30-feet long corridor located at the palliative care unit.

Resistance exercise: Patient is assessed for the ability to use 1lb of dumbbell, if they are able to use easily then he has to use 2lb dumbbell. Dumbbell exercises during the first week are 10 repetitions, which will increase 10 repetitions per week, reaching a total of 40 repetitions on the last week. The exercises will be:

1. - shoulder flexion 0-180º;
2. - shoulder abduction and adduction;
3. - shoulder extension;
4. - elbow flexion;
5. - wrist flexion and extension;

Patients' will have monitored their blood pressure, heart/cardiac frequency ( 40-60% of HR RESERVE or 60-70% HR MAX) and oxygen saturation by way of a finger oximeter made by Digit and perceived effort = light sweating, increase HR and breathing. Daily walk in the Borg scale at the beginning, middle and end will be applied to evaluate the fatigue of the patient.

ELIGIBILITY:
Inclusion Criteria:

* Be older than 18 years of age,
* Any gender
* Able to understand the study protocol,
* Functional capacity equal to or higher than 60, according to the Karnofsky scale,
* Patients with a life expectancy between 3 and 12 months,
* Patient able to ambulate independently without need for any orthotics.

Exclusion Criteria:

* Patients that use drugs in order to control fatigue (Methylphenidate, Modafinil),
* Anemic Patients (HB< 8.0 mg/dl),
* Patients with cognitive deficit,
* Uncontrolled pain higher than 5, according to Visual Analogue Scale (VAS),
* Patients currently exercising,
* Patients with congestive heart failure (CHF) (New York Heart Association functional class III or IV) or related angina.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-12; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Fatigue | Baseline, 7 days, 14 days and 20 days after starting the intervention.
  ESAS score and FACT-F questionnaire.

SECONDARY OUTCOMES:
Quality of life | Baseline, 7 days, 14 days and 20 days after starting the intervention.
  EORTC QLQ-C30.
Anxiety and Depression Evaluation | Baseline, 7 days, 14 days and 20 days after starting the intervention.
  Anxiety & Depression Hospital Anxiety Depression scale (HADS)
Patient impression satisfaction | Baseline and 7 days after starting the intervention
  Satisfaction-PGIC.

CONTACTS AND LOCATIONS:
Overall Officials: Adriana M Ferreira, PhD, Principal Investigator — Barretos Cancer Hospital
Locations (1):
- São Judas Tadeu Hospital, Barretos, São Paulo, Brazil